CLINICAL TRIAL: NCT00358267
Title: A Randomized Trial Comparing Two Surgical Techniques for Inferior Turbinate Reduction
Brief Title: Randomized Trial Comparing Partial Resection of Inferior Turbinate(PRIT) and Radiofrequency Ablation(RFA) for Inferior Turbinate Reduction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Michael G. Stewart MD MPH, Weill Medical College of Cornell University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0603008446
Record Dates: First submitted 2006-07-27; First posted 2006-07-31 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Nasal Obstruction; Septal Deformity; Turbinate Hypertrophy
Keywords: Inferior Turbinate Reduction; Partial Resection of Inferior Turbinates (PRIT); Radiofrequency Ablation (RFA); NOSE scale; Nasal Obstruction
MeSH Terms: conditions — Nasal Obstruction | interventions — Radiofrequency Ablation

ARMS (2):
- RFA (Active Comparator): Radiofrequency Ablation (RFA) involves inserting a special needle into the inferior (lower) turbinate that releases high frequency energy, which produces heat. The energy and heat cause tissue denaturation (protein damage) and vaporization. The vaporization reduces tissue volume, and denaturation causes healing with scar tissue formation and contraction of surrounding tissue. This procedure can be done under local anesthesia at the doctor's office.
  Interventions: Procedure: Radiofrequency Ablation (RFA)
- PRIT (Active Comparator): Partial Resection of Inferior Turbinate (PRIT) involves surgically removing a small piece off the turbinate, which also reduces its size.
  Interventions: Procedure: Partial Resection of Inferior Turbinates (PRIT)

INTERVENTIONS:
Procedure: Partial Resection of Inferior Turbinates (PRIT) — PRIT involves surgically removing a small piece off the turbinate, which also reduces its size.
  Arms: PRIT
Procedure: Radiofrequency Ablation (RFA) — RFA involves inserting a special needle into the inferior (lower) turbinate that releases high frequency energy, which produces heat. The energy and heat cause tissue denaturation (protein damage) and vaporization. The vaporization reduces tissue volume, and denaturation causes healing with scar tissue formation and contraction of surrounding tissue. This procedure can be done under local anesthesia at the doctor's office.
  Arms: RFA

SUMMARY:
Turbinates are large structures in the nasal airway that help the nose to clean and humidify the air we breathe. Inferior turbinates can swell up and block the breathing passage, making it hard to breath. To address this, turbinate size must be reduced.

This study looks at two common procedures for turbinate reduction:

1. Radiofrequency Ablation (RFA) involves inserting a special needle into the inferior (lower) turbinate that releases thermal energy, which significantly reduces its size. This can be done under local anesthesia at the doctor's office.
2. Partial Resection of Inferior Turbinate (PRIT) involves surgically removing a piece off the turbinate, which also reduces its size.

While both procedures improve nasal obstruction, no study has directly compared which is more effective.

Eighty patients being treated for septal deformity and turbinate hypertrophy will be randomly chosen for either PRIT or RFA treatment. They will fill out a simple, five question survey that measures how they view their nasal blockage 4 times in one year. We believe that since PRIT permanently removes a part of the turbinate, PRIT patients will report more improvement than RFA patients one year later. We believe that complications (measured by the doctor) will be the same for both treatments.

DETAILED DESCRIPTION:
Subjective nasal obstruction is usually caused by intranasal anatomic obstruction. A critical area is the anterior nasal valve, and nasal septal deformity and inferior turbinate hypertrophy often combine to produce symptomatic obstruction at the anterior valve.

Surgical treatments to reduce turbinate size and also to correct nasal septal deformity have been shown to be effective at improving nasal obstruction. While many studies have demonstrated the improvements after surgery, most prior studies assessed outcome using non-validated questionnaires, or primitive measures such as a single-item rating scale.

There is now a validated, patient-based, outcome instrument to assess nasal obstruction, which is valid, reliable, and sensitive: the Nasal Obstruction Symptom Evaluation (NOSE) scale (Stewart, Witsell, et al). This brief and easy to complete instrument is a valid measure of the patient's perception of nasal obstruction. A multi-center prospective study using the NOSE scale showed that septoplasty alone resulted in significant improvement in nasal obstruction, and septoplasty with PRIT had an even larger improvement in nasal obstruction, although the difference did not reach statistical significance because of sample size (Stewart, Smith, et al). Nevertheless, turbinate reduction appeared to have some additive effect on symptomatic improvement, which is a clinical findings that has been noted by surgeons for many years.

The techniques of inferior turbinectomy have evolved over time. Initially, partial or even total resection of the inferior turbinate was performed. However, total inferior turbinate resection was found to have a high rate of several long-term complications, including excessive dryness (rhinitis sicca), atrophic rhinitis, crusting, bleeding, etc. (Moore GF, Moore EJ), and this technique is generally not performed today. By extension, many surgeons have been concerned about the potential sequelae of partial inferior turbinectomy, even though large prospective series have demonstrated excellent outcomes and minimal complications from the PRIT technique (Fanous, Ophir, Grymer, Stewart/Smith).

Several alternative techniques for turbinate volume reduction - that do not involve full-thickness resection of a portion of the turbinate - have been reported, and all seem to be effective in single-modality series (Nease, Bhattacharyya, Utley, Li). In fact, anecdotally many surgeons claim that RFA is as effective as PRIT. In addition, radiofrequency techniques can be performed under local anesthesia in the office setting, which increases the ease of use. While RFA is appealing because it can be performed under local anesthesia, the improved ease of use must be weighed against the potential for lower effectiveness, since tissue is not removed. There are no data from direct comparative studies, probably partly because there has not been a validated outcome tool available.

Therefore, sufficient clinical equipoise exists to randomize patients to receive one of these two widely-accepted techniques.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects will be male or female, 18 years or older, with nasal septal deformity and bilateral inferior turbinate hypertrophy

Exclusion Criteria:

* Subjects with contraindication to general anesthesia or nasal surgery
* Additional simultaneous nasal surgery, such as sinus surgery or rhinoplasty
* Nasal polyposis and prior inferior turbinectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoint for the 80 subjects enrolled will be the NOSE Score at 12 months. | 12 months

SECONDARY OUTCOMES:
The prevalence of complications. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Stewart, MD, MPH, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

REFERENCES:
- [Background] Nease CJ, Krempl GA. Radiofrequency treatment of turbinate hypertrophy: a randomized, blinded, placebo-controlled clinical trial. Otolaryngol Head Neck Surg. 2004 Mar;130(3):291-9. doi: 10.1016/j.otohns.2003.11.003. PMID 15054369
- [Background] Bhattacharyya N, Kepnes LJ. Clinical effectiveness of coblation inferior turbinate reduction. Otolaryngol Head Neck Surg. 2003 Oct;129(4):365-71. doi: 10.1016/S0194-59980300634-X. PMID 14574290
- [Background] Grymer LF, Illum P, Hilberg O. Septoplasty and compensatory inferior turbinate hypertrophy: a randomized study evaluated by acoustic rhinometry. J Laryngol Otol. 1993 May;107(5):413-7. doi: 10.1017/s0022215100123308. PMID 8326220
- [Background] Ophir D, Schindel D, Halperin D, Marshak G. Long-term follow-up of the effectiveness and safety of inferior turbinectomy. Plast Reconstr Surg. 1992 Dec;90(6):980-4; discussion 985-7. PMID 1448533
- [Background] Moore GF, Freeman TJ, Ogren FP, Yonkers AJ. Extended follow-up of total inferior turbinate resection for relief of chronic nasal obstruction. Laryngoscope. 1985 Sep;95(9 Pt 1):1095-9. PMID 4033334
- [Background] Fanous N. Anterior turbinectomy. A new surgical approach to turbinate hypertrophy: a review of 220 cases. Arch Otolaryngol Head Neck Surg. 1986 Aug;112(8):850-2. doi: 10.1001/archotol.1986.03780080050010. PMID 3718689
- [Background] Moore EJ, Kern EB. Atrophic rhinitis: a review of 242 cases. Am J Rhinol. 2001 Nov-Dec;15(6):355-61. PMID 11777241
- [Background] Stewart MG, Smith TL, Weaver EM, Witsell DL, Yueh B, Hannley MT, Johnson JT. Outcomes after nasal septoplasty: results from the Nasal Obstruction Septoplasty Effectiveness (NOSE) study. Otolaryngol Head Neck Surg. 2004 Mar;130(3):283-90. doi: 10.1016/j.otohns.2003.12.004. PMID 15054368
- [Background] Stewart MG, Witsell DL, Smith TL, Weaver EM, Yueh B, Hannley MT. Development and validation of the Nasal Obstruction Symptom Evaluation (NOSE) scale. Otolaryngol Head Neck Surg. 2004 Feb;130(2):157-63. doi: 10.1016/j.otohns.2003.09.016. PMID 14990910
- [Background] Utley DS, Goode RL, Hakim I. Radiofrequency energy tissue ablation for the treatment of nasal obstruction secondary to turbinate hypertrophy. Laryngoscope. 1999 May;109(5):683-6. doi: 10.1097/00005537-199905000-00001. PMID 10334213
- [Background] Li KK, Powell NB, Riley RW, Troell RJ, Guilleminault C. Radiofrequency volumetric tissue reduction for treatment of turbinate hypertrophy: a pilot study. Otolaryngol Head Neck Surg. 1998 Dec;119(6):569-73. doi: 10.1016/S0194-5998(98)70013-0. PMID 9852527